CLINICAL TRIAL: NCT04487275
Title: MLC901 for Moderate to Severe Traumatic Brain Injury: Pilot, Randomized, Double-Masked, Placebo-controlled Trial
Brief Title: MLC901 for Moderate to Severe Traumatic Brain Injury (Specified Drug Code)
Acronym: MLC901
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ali Amini Harandi (Other)
Responsible Party: Sponsor-Investigator, Ali Amini Harandi, Prof, Shahid Beheshti University
Organization: Shahid Beheshti University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-299
Record Dates: First submitted 2020-07-17; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Neuroaid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug (Experimental): MLC901 capsules three times per day over 6 months
  Interventions: Drug: MLC901 or Placebo
- Placebo (Placebo Comparator): Placebo capsules three times per day over 6 months
  Interventions: Drug: MLC901 or Placebo

INTERVENTIONS:
Drug: MLC901 or Placebo — groups randomly assigned to receive either MLC901 or placebo capsules three times per day over 6 months
  Other Names: Placebo

SUMMARY:
Patients with a diagnosis of moderate to severe traumatic brain injury (TBI) will be enrolled. Subjects will be randomly assigned to receive either MLC901 (Specified Drug Code) or placebo capsules three times per day over 6 months. Evaluation of patients will be carried out at baseline as well as at 3-month and 6-month follow-up visits. Modified Rankin Scale (mRS) and Glasgow outcome scale (GOS) will be used to examine patients. Efficacy will be evaluated by comparing these two scores between the 2 groups at follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* age between 15 and 65
* non-penetrating moderate (Glasgow Coma Scale score [GCS] 9-12) or severe (GCS 3-8) traumatic brain
* injury less than 24 hrs from traumatic injury
* anticipated intensive care unit length of stay at least 48 hrs

Exclusion Criteria:

* GCS = 3 and fixed dilated pupils or penetrating injury
* coexisting injury or medical conditions which could adversely affect our study outcome measures
* dependence for everyday activities before the injury
* pregnancy or breastfeeding
* known allergy to any of MLC901 components

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-08-20 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
functional outcome 1 | at baseline
  functional outcome scales of GOS
functional outcome 2 | at 3rd month post-injury
  functional outcome scales of GOS
functional outcome 3 | at 6th month post-injury
  functional outcome scales of GOS
functional outcome 4 | at baseline
  functional outcome scales of MRS
functional outcome 5 | at 3rd month post-injury
  functional outcome scales of MRS
functional outcome 6 | at 6th month post-injury
  functional outcome scales of MRS

CONTACTS AND LOCATIONS:
Locations (1):
- Brain Mapping Research Center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided